CLINICAL TRIAL: NCT05547048
Title: Integrated eHealth for HIV and Substance Use Disorders in Justice Involved Women
Brief Title: Integrated e-Health (Electronic Health) for HIV and Substance Use Disorders in Justice Involved Women
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000033006; 1R01DA057342-01 (NIH)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: HIV; Opioid Use Disorder; eHealth
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: This study will compare the Athena strategy to a decision aid-only intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Athena Strategy (Experimental): Virtual care model that includes direct synchronous videoconferencing with a provider, telephone/ texting communication, electronic health records, e-prescribing for the purposes of delivering PrEP and medications for opioid use disorder. This is combined with a decision aid for PrEP
  Interventions: Combination Product: Athena strategy
- Decision Aid (Active Comparator): Decision aid for PrEP tailored for justice-involved women with opioid use disorder
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — Decision aid for PrEP tailored for justice-involved women with opioid use disorder
  Arms: Decision Aid
Combination Product: Athena strategy — eHealth for integrated PrEP/medications for opioid use disorder + decision aid
  Arms: Athena Strategy

SUMMARY:
The purpose of this 2-site (CT, AL) study is to test innovative interventions to reduce stigma and improve the pre-exposure prophylaxis (PrEP) and opioid use disorder (OUD) care continua in women involved in the criminal justice system (WICJ).

This study evaluates a newly validated PrEP decision aid and eHealth for integrated PrEP and MOUD compared to a decision aid-only for WICJ with OUD.

DETAILED DESCRIPTION:
Problem: There is urgent need to reach women involved in criminal justice (WICJ) for lifesaving, evidence-based PrEP and medications for OUD (MOUD), using innovative healthcare delivery models that surmount existing social and structural barriers to engagement.

Purpose: This study uses a newly validated decision aid and eHealth to remotely deliver integrated PrEP and MOUD to community-based WICJ with OUD in New Haven, Connecticut (CT) and Birmingham, Alabama (AL).

Methods: 250 PrEP-eligible WICJ with OUD will undergo randomization to: a) the "Athena" strategy, which includes the decision aid + eHealth for remote integrated PrEP/MOUD with a provider using outputs from the decision aid; or b) decision aid-only with referral to community-based PrEP/MOUD. Randomization will be stratified by site; past 6-month use of any stimulants; and baseline receipt of MOUD. Follow-up study assessments occur at months 1, 3, and 6. To understand implementation, the investigators will conduct population modeling and engage with relevant stakeholders through focus groups using nominal group technique and in-depth individual interviews.

Aims: The Aims of the project are: 1) To compare the Athena strategy to decision aid-only in terms of patient-level engagement in the PrEP and OUD care continua, considering key site differences; and 2) To assess scale-up potential of the Athena strategy in terms of modelled long-term outcomes and how stakeholders interact with eHealth for integrated PrEP/MOUD in WICJ in two diverse epidemiological and implementation contexts (CT and AL), using standardized definitions of implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* cis-women
* have access to a working mobile or landline phone
* Lifetime CJ-involvement (probation, parole, intensive pretrial or community supervision, or release from prison/jail)
* are confirmed HIV-negative by point-of-care 3rd generation HIV antibody test
* meet clinical criteria for PrEP
* have opioid use disorder (regardless of baseline treatment status)

Exclusion Criteria:

* unable or unwilling to provide informed consent
* pregnant or breast-feeding
* currently taking PrEP at the time of study enrollment
* not comfortable conversing in English or Spanish.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who initiate PrEP | up to 6 months
  PrEP in initiation will be determined using dates of prescription and pharmacy fill and medication type (brand/generic)

SECONDARY OUTCOMES:
Number of participants who are adherent to PrEP | up to 6 months
  PrEP adherence will be assessed using a urine assay for measuring tenofovir levels (single point of care qualitative immunoassay reflecting past 48-hour adherence), where a positive test results indicates adherence.
Number of participants who engage in opioid use disorder treatment | up to 6 months
  The opioid use disorder treatment cascade engagement is composed of and defined by: 1) initiation of medications for opioid use disorder (or other evidence-based treatment); 2) 6-month retention on treatment; and 3) remission. The study will assess for complexity of substance use disorder treatment (e.g., court mandated vs. voluntary, behavioral vs. MOUD, residential vs. outpatient, detoxification program, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Price, MPA, Study Director — Yale University; Jaimie P Meyer, MD, MS, FACP, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - University of Alabama in Birmingham, Birmingham, Alabama
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer JP, Brunson S, Price CR, Mulrain M, Nguyen J, Altice FL, Kyriakides TC, Cropsey K, Eaton E. Rationale and design of a randomized clinical trial of integrated eHealth for PrEP and medications for opioid use disorders for women in the criminal legal system. The Athena study. Addict Sci Clin Pract. 2025 Jan 17;20(1):4. doi: 10.1186/s13722-024-00534-x. PMID 39825419